CLINICAL TRIAL: NCT05692921
Title: Tailoring Post Discharge (TPD) - Bridging the Gap Through Education and Community Support
Brief Title: Tailoring Post Discharge (The TPD Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Shuangbo Liu, Principal Investigator, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TPD Protocol
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: Percutaneous Coronary Intervention; Education; Community Support; Remote Home Monitoring; Rapid Response Nurses; Low-risk assessment
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Comparing 2 interventional groups: 1) Virtual Remote Home Monitoring and 2) Rapid Response Nursing care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote Home Monitoring (RHM) (Experimental): Remote Home Monitoring Platform (RHM): will be utilized to help tailor education and support for the patient after they have been discharged from the hospital. The platform will provide access to and delivery of health related education and information for continued self-care within the community. The platform will be used to evaluate post discharge symptoms and for health care providers to access the need for continued direct patient care and education through virtual processes.
  Interventions: Other: Remote Home Monitoring (RHM)
- Rapid Response Nursing (RRN) (Active Comparator): Rapid Response Nursing Team (RRN): The RRN will help clients/patients to:
  * Understand their current health conditions, treatments, how to manage symptoms and when/who to ask for help; Specifically; they will
  * Help clients to understand their hospital discharge plan;
  * Support patients during their recovery at home;
  * Reinforce and contribute to in-hospital education about heath health and recovering safely at home;
  * Review medications to help clients understand the purpose, side effects and how to take prescribed medications correctly, including assisting clients with getting prescriptions filled;
  * Connect with their Home Clinic, ensuring everyone has the necessary information for follow-up care;
  * Connect clients with a Home Clinic if they do not have one; and
  * Access appropriate home supports to help clients remain at home safely for as long as possible.
  Interventions: Other: Rapid Response Nursing
- Registry (No Intervention): Registry Arm:
  Patients who fit the criteria for study inclusion and choose not to participate in the main study will be provided with an opportunity to consent to the registry arm of the study. The registry arm of the study is an opportunity to establish a standard of care group free from research bias. Patients who enroll in the registry will only need to complete a short questionnaire before they are discharged home which will take approximately 5 minutes. Additionally, research staff will also complete a medical chart review to identify specific medical information related to their demographics, cardiac procedure, hospital stay, recovery, and to identify any re-admissions to hospital that may have occurred after the patient has been discharged home.

INTERVENTIONS:
Other: Remote Home Monitoring (RHM) — A Virtual platform will be used to provide education and support for ACS patients within the community after a patient is discharged home
  Arms: Remote Home Monitoring (RHM)
Other: Rapid Response Nursing — A Rapid Response Nurse will be used to provide education and support for ACS patients within the community after a patient is discharged home.
  Arms: Rapid Response Nursing (RRN)

SUMMARY:
This randomized control trial seeks to better understand the educational needs of Acute Coronary Symptom (ACS) patients including the optimal timing and method of delivery as well as linkages with appropriate community resources and supports are important for cardiac patients to self-manage post hospital discharge to improve outcomes. While there is some literature of the learning needs of ACS patients, there is a paucity of research related to the timing and preferred methods of delivery. This study aims to better understand how best to tailor care for ACS patients from hospital to community. Specifically, the investigators propose a 2 phased approach to understand the needs of patients, and then to develop and deliver a tailored approach to assess, educate and support patients both in-hospital and within the community. The intervention compares 1) a virtual remote home monitoring (RHM) platform and 2) Rapid Response Nursing (RRN) staff to follow, educate and support ACS patients post hospital discharge for a period of no more than 30 days.

The Primary Objective of this study is to safely transition low risk ACS patients, from hospital to home, with appropriate supports to safely self-manage in the community and to provide educational and community supports to improve post discharge outcomes of low risk ACS patients

DETAILED DESCRIPTION:
Study design: 2 phase single center randomized, prospective pilot study

Phase 1) Evaluation of quality indicator results from discharge questionnaires from patients post ACS and a further investigation through patient engagement techniques about education, community support and quality of care. This process, comprising of patient collaborators/partners, will contribute to the study design, tool and resource development.

Phase 2) Randomized trial - Intervention (low risk 24-hour discharge support using Rapid Response nursing (RRN) vs low risk 24-hour discharge support using Remote Home Monitoring (RHM). Patients will be assessed using a trialed multipoint tool developed for this research study utilizing the cardiac, medical, community and patient risks. After assessment, low-risk patients will be randomized into the study. The study interventions will utilize either the RRN or the RHM to deliver education and support to patients post discharge.

Phase 1 - Patient Engagement Panel:

Patient engagement in research involves meaningful and active collaboration between patients and researchers throughout the different phases of a research project, including planning, data collection, data analysis, and knowledge translation. These collaborative meetings inform and guide study development. The central tenet of patient engagement in research is that, while clinicians and investigators have disease and research specific expertise, patients have expertise that stems from lived experience of their health issues. By sharing their experiences of the daily impact of disease and their perspectives regarding unmet needs, therapeutic burdens, balance of benefits and risks, and types of research questions most important to them, patients can transform the research process from one directed by investigators to one driven and informed by the needs of patients and their caregivers.

To generate information to refine the implementation plan of the study the investigators intend to recruit individuals to our Patient engagement panel who previously had ACS care and hospitalization at the St. Boniface Hospital and/or caregivers for the ACS patient. The investigators will construct panel members that reflect key demographic characteristics of our study's target population (including age, sex, gender, rural vs urban home location, and type of ACS) and other relevant selection criteria. These engagement activities will look to provide valuable insight into their experiences, while in-hospital and their transition back to the community, to help us develop patient centered education and post-discharge support. The investigators expect to generate patient and caregiver knowledge over 3 sessions within a 2-week period of time. Each session will be approximately 2 hours in length and will be mediated by research staff who have extensive experience in patient engagement. These sessions will either be in person or virtual, which will be dependent on participant needs.

From the patient engagement panel, The investigators will select 2 participants to become patient collaborators with our research team. These patients will provide information to help guide the refinement of study design, study procedures (e.g., recruitment methods, approaches to maximize education retention, use of accessible language in recruitment and study materials, and usability of technology), relevance of outcomes to patient concerns, data analysis (e.g., interpretation and contextualization of findings), and knowledge translation (e.g., alternate dissemination methods, use of accessible language, manuscript development). The anticipated lifespan of this patient- collaborators participation is from study planning through to the end of study knowledge translation (approximately 2 years) consisting of formal and informal meetings during this time period.

Phase 2 - Prospective Research:

Main Study Participants:After a successful PCI and assessing patients' risk criteria, patients who are considered low risk will be identified by the attending cardiology staff. Research staff will then be provided the names of these patients and they will then approach the patient for consent, prior to hospital discharge. Patients, upon consenting to the study, will be provided several questionnaires to complete and then randomized to one of two arms, the RRN arm or the RHM arm.

Low Risk Assessment Process (Hybrid):

The cardiology team at the St. Boniface Hospital will first utilize the Zwolle (STEMI) or the Grace (NSTEMI) scores to initially assess low medical risk for ACS patients. Both scores have been previously validated. 3-5 As many as 30 additional factors will be considered when completing the scoring for low-risk inclusion (Appendix 1). These factors include social, economic, cognitive, mental and physical dimensions.

Randomization:

Utilizing an online randomization tool (www.HTTPS//randomizer.org) participants who consent to the main study are assigned to either RRN intervention arm or the RHM intervention arm in a blocked 1:1 format.

Registry Participants Patients who fit the criteria for study inclusion and choose not to participate in the main study will be provided with an opportunity to consent to the registry arm of the study. The registry arm of the study is an opportunity to establish a standard of care group free from research bias. Patients who enroll in the registry will only need to complete a short questionnaire before they are discharged home which will take approximately 5 minutes. Additionally, research staff will also complete a medical chart review to identify specific medical information related to their demographics, cardiac procedure, hospital stay, recovery, and to identify any re-admissions to hospital that may have occurred after the patient has been discharged home.

Standard of Care:

Currently, education is delivered by several health care providers, including Nursing, Occupation and Physical Therapy, Pharmacy, Dieticians and Physicians. Delivery of the education material vary based on availability of health care providers and the length of time a patient is admitted to the hospital as well as timing of discharge (weekday vs weekend). Patients are discharged with educational material such as: Heart and Stroke's "Living well with Hearts Disease" booklet, information on Coronary angiograms and angioplasty/stents, and medication information sheets provided by pharmacy. A clinical decision is made by the health care team regarding whether the patient needs cardiology follow up. While most STEMI patients are referred to a cardiologist (if they don't already have one), the practice is variable for NSTEMI and unstable angina patients. This standard of care will continue to be provided to all ACS patients being discharged from the St. Boniface Hospital.

Intervention:

Education Development and Implementation:

Focused and adaptable educational material will be created to support the patients upon hospital discharge. This education and support component will either be administered by the Rapid Response Nurses (RRN) who will be delivering, in person or virtually, or the Remote Home Monitoring (RHM) system delivered virtually. Instead of routine education for all patients, through this intervention, the appropriate education will be provided at the appropriate time for patients based on their own learning needs. The existing educational material will be revised to be more digestible and using multiple methods of learning, including infographics, education, short summaries, etc. The education will be developed in coordination with patient and clinical teams. Further work throughout the patient engagement phase 1 needs to:

* Provide directed and tailored education (publication and access to electronic documents) and community support, based on patient engagement sessions and current health care directives.
* Evaluate all discharge resource material
* understand current content and process
* identify and integrate changes
* Identify community supports available for post ACS patients
* Create resource sheet
* Engage community partners
* Cardiac Rehabilitation (CR) facilities
* Community health care support (i.e. access centres)

Rapid Response Nursing Team:

The RRNs will meet with study participants on 3 occasions. 1) 24 hours post hospital discharge, 2) 5-7 days post hospital discharge, and 3) 2-week post hospital discharge. While the initial visit will be in person, the next two visits may be in person or virtual (phone/tablet/computer) depending on patient preference. The RRN will help clients/patients to:

* Understand their current health conditions, treatments, how to manage symptoms and when/who to ask for help; Specifically; they will
* Help clients to understand their hospital discharge plan;
* Support patients during their recovery at home;
* Reinforce and contribute to in-hospital education about heath health and recovering safely at home;
* Review medications to help clients understand the purpose, side effects and how to take prescribed medications correctly, including assisting clients with getting prescriptions filled;
* Connect with their Home Clinic, ensuring everyone has the necessary information for follow-up care;
* Connect clients with a Home Clinic if they do not have one; and
* Access appropriate home supports to help clients remain at home safely for as long as possible.

Remote Home Monitoring Platform:

* The remote home monitoring platform will be utilized to help tailor the education and support for the patient.
* Engage patients
* Providing access to and delivery of health related education and information for continued self-care within the community.
* Evaluating post discharge symptoms
* Algorithm to define and deliver continued patient care throughout the "at home recovery process" - green, yellow, and red flag system
* Accessibility by health care provider to assess the need for continued direct patient care and education
* Delivery of surveys for research purposes
* Patients will be provided access to this platform on their own device, whether mobile phone, tablet or home computer.
* If the patient does not have access to this technology a tablet will be provided to the patient for the purposes and duration of this research study.
* There is no cost to the patient for this.
* This system has been approved and adopted by shared health for the remote home monitoring of patients after they have been discharged home from the hospital

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who presented with ACS to St. Boniface Hospital
* Considered low risk based on cardiac risk, comorbidities, community and patient resources

Exclusion Criteria:

* Age less than 18 years.
* Unable or unwilling to provide consent
* Considered high risk for early discharge
* Lives outside of Winnipeg (for Phase 2 of the study, we will only be focusing on patients that live within Winnipeg)
* No internet or mobile data access

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Mortality - Composite outcome measure | 30-days post hospital discharge
  mortality - measured as yes/no (Alive at 30 days = no)
Repeat MI - Composite outcome measure | 30-days post hospital discharge
  repeat myocardial infarction - measured as yes/no (repeat MI at 30 days = yes)
Re-Admission - Composite outcome measure | 30-days post hospital discharge
  re-hospitalization and emergency room/urgent care visits measured as yes/no (rehospitalization at 30 days = yes)
Congestive Heart Failure - Composite outcome measure | 30-days post hospital discharge
  congestive heart failure - measured as yes/no (Ejection fraction < 40% is CHF)
Congestive Heart Failure - Composite outcome measure | 30-days post hospital discharge
  serious arrhythmia (VT, VF) measured as yes/no (Arrhythmia at 30 days = yes)

SECONDARY OUTCOMES:
EQ-5D-5L - Health related Quality of Life | baseline (before discharge from hospital), 2-weeks post hospital discharge, and 30 Days post hospital Discharge
  EQ-5D-5L - This survey will measure 5 aspects of self-reported quality of life for patients. Each component is scored from 1-5 with a total score of the tool from 5-25. Lower scores indicate better outcomes
EQ-VAS - Health related Quality of Life | baseline (before discharge from hospital), 2-weeks post hospital discharge, and 30 Days post hospital Discharge
  EQ-VAS - this survey measures self-report quality of life on a scale of 0-100 Higher scores indicate better self reported Quality of life
General Anxiety Disorder (GAD) - 7 | baseline (before discharge from hospital), 2-weeks post hospital discharge, and 30 Days post hospital Discharge
  GAD-7 this survey measures self-report anxiety symptoms with a total score from 0-21. Lower scores indicate fewer anxiety symptoms
Patient Health Questionnaire (PHQ) - 9 | baseline (before discharge from hospital), 2-weeks post hospital discharge, and 30 Days post hospital Discharge
  PHQ-9 this survey measures self-report depression symptoms with a total score from 0-27. Lower scores indicate fewer depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada